CLINICAL TRIAL: NCT04107805
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Rising Oral Doses of BI 1323495 Versus Placebo in Healthy Subjects, Including an Investigation of Drug-drug Interaction With Microdose Midazolam (Double-blind, Randomised, Placebo-controlled [Within Dose Groups] Trial)
Brief Title: A Study in Healthy Men and Women to Test How Well Different Doses of BI 1323495 Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 1405-0002; 2018-004238-13 (EudraCT Number)
Record Dates: First submitted 2019-09-26; First posted 2019-09-27 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- 10 mg BI 1323495 bid EM (Experimental)
  Interventions: Drug: BI 1323495
- 10 mg BI 1323495 bid PM (Experimental)
  Interventions: Drug: BI 1323495
- 30 mg BI 1323495 bid EM (Experimental)
  Interventions: Drug: BI 1323495
- 30 mg BI 1323495 bid PM (Experimental)
  Interventions: Drug: BI 1323495
- 70 mg BI 1323495 bid + Midazolam EM (Experimental)
  Interventions: Drug: BI 1323495; Drug: Midazolam
- 120 mg BI 1323495 bid + Midazolam EM (Experimental)
  Interventions: Drug: BI 1323495; Drug: Midazolam
- 120 mg BI 1323495 qd EM (Experimental)
  Interventions: Drug: BI 1323495
- 150 mg BI 1323495 bid + Midazolam EM (Experimental)
  Interventions: Drug: BI 1323495; Drug: Midazolam
- Placebo/Placebo+ Midazolam (Experimental)
  Interventions: Drug: Placebo; Drug: Midazolam

INTERVENTIONS:
Drug: BI 1323495 — Tablet
  Arms: 10 mg BI 1323495 bid EM; 10 mg BI 1323495 bid PM; 120 mg BI 1323495 bid + Midazolam EM; 120 mg BI 1323495 qd EM; 150 mg BI 1323495 bid + Midazolam EM; 30 mg BI 1323495 bid EM; 30 mg BI 1323495 bid PM; 70 mg BI 1323495 bid + Midazolam EM
Drug: Placebo — Tablet
  Arms: Placebo/Placebo+ Midazolam
Drug: Midazolam — Oral administration
  Arms: 120 mg BI 1323495 bid + Midazolam EM; 150 mg BI 1323495 bid + Midazolam EM; 70 mg BI 1323495 bid + Midazolam EM; Placebo/Placebo+ Midazolam

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 1323495 in healthy subjects following bid oral administration of multiple rising doses, each over an 11 day treatment period.

Secondary objectives are the exploration of the pharmacokinetics (PK) including dose proportionality (only for Part 1) as well as attainment of steady state. This includes exploration of a therapeutic exposure range, a range not adequately achieved in the single-rising dose trial 1405-0001.

ELIGIBILITY:
Inclusion criteria:

* Healthy subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), PR), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 70 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* For Part I: Subjects genotyped as UGT2B17 extensive metabolizers, i.e., carrying at least one functional allele of the UGT2B17 gene (*1/*1 or *1/*2).

For Part II: Subjects genotyped as UGT2B17 poor metabolizers, i.e., carrying no functional allele of the UGT2B17 gene (*2/*2)

-Male or female subjects:

* For 'female subjects not of childbearing potential' at least one of the following criteria must be fulfilled:
* Permanently sterile (permanent sterilisation methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy)
* Postmenopausal, defined as at least 1 year of spontaneous amenorrhea without an alternative medical cause (in questionable cases a blood sample with FSH above 40 U/L and estradiol below 30 ng/L is confirmatory)
* Female subjects of childbearing potential must use a highly effective contraception method from at least 30 days before the first administration of trial medication until 14 days after trial completion

Exclusion criteria:

* Any finding in the medical examination (including Blood Pressure (BP), PR, or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator. In particular a marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) at screening
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance; safety laboratory screening evaluation can be repeated a maximum of two times
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator or at risk of requiring concomitant drug therapy, e.g., gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorder, diseases of the central nervous system (including, but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients); mild seasonal allergy adequately managed by topic administration of drugs to eyes or nose is not excluded
* Subjects with a documented active malignancy, or malignancy for which the subject has undergone resection, radiation therapy, or drug therapy (e.g., cytostatic, protein kinase inhibitor, or immune checkpoint inhibitor therapy), within the last 5 years.
* Subjects who have been previously randomised in this study.
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days, or within 5 half-lives of the investigational drug (whichever is longer), of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Major surgery (major according to the investigator's assessment) performed within 6 weeks prior to randomisation or planned within 3 months after screening, e.g. hip replacement.
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day), also inability to refrain from smoking during in-house confinement
* Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males) or any other drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subjects with veins unsuited for venipuncture (for instance, veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture) as assessed by the investigator.
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male subjects with 'women of childbearing potential' (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after the last administration of trial medication
* Known relevant immunodeficiency, as judged by the investigator
* Chronic or relevant acute infections
* History and/or presence of tuberculosis; positive result for interferon gamma release assay (IGRA) (i.e., QuantiFERON TB-Gold), or history of pneumococcal infection
* Positive results for Hepatitis B antigen, Hepatitis C antibodies, and/or human immunodeficiency virus (HIV) 1 antigen or HIV1/2 antibodies, at screening
* Aural body temperature of more than 37.7°C on Day -3 to -1, or Day -4 to -2 for subjects receiving Midazolam microdosing.
* Subjects who have received live or live-attenuated vaccine in the 4 weeks prior to dosing
* C-reactive protein above upper limit of laboratory reference range at screening and/or on Day -3 to -1, or Day -4 to -2 for subjects receiving Midazolam microdosing.
* Subjects with signs of current gingivitis/periodontitis. Inspection of the oral cavity will be performed by the investigator.
* Current or history of relevant kidney, urinary tract diseases or abnormalities (e.g. nephrolithiasis, hydronephrosis, acute or chronic nephritis, renal injury, renal failure), according to investigator.
* Estimated glomerular filtration rate (eGFR) according to CKD-EPI formula < 80 mL/min at screening.
* Known clinically relevant impairment of liver function or clinically relevant laboratory abnormality at the screening visit (V1) regarding liver aminotransferases, alkaline phosphatase, gamma glutamyl transferase, bilirubin, serum albumin, as judged by the investigator.
* Subjects with a known coagulopathy or abnormal coagulation laboratory parameters at screening, or subjects who, within 10 days prior to administration of trial medication, used any drug that could reasonably inhibit coagulation
* Females with a positive pregnancy test or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fraunhofer ITEM, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a trial to assess safety, tolerability, pharmacokinetics, and pharmacodynamics of multiple rising oral doses of BI 1323495 versus placebo in healthy subjects, including an investigation of drug-drug interaction with microdose midazolam (double-blind, randomised, placebo-controlled [within dose groups] trial).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo/Placebo + Midazolam: This arm comprises placebo only treated participants and those participants who received placebo + midazolam. Placebo only treated participants were administered film-coated tablets of placebo matching BI 1323495 dosage and participants who received placebo + midazolam were administered film-coated tablets of placebo matching BI 1323495 dosage + a single daily dose of 1.5 milliliter (mL) of solution for injection of midazolam concentrated 50 microgram (ug)/mL (total dosage=75 ug) orally with 240 mL of water within 30 minutes after a standard breakfast on Day -1 and on Day 11.
- 10 mg BI 1323495 Bid EM: Participants carrying at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) one film-coated tablet of 10 milligram (mg) of BI 1323495 orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal.
- 10 mg BI 1323495 Bid PM: Participants carrying no functional allele of the UGT2B17 gene (poor metabolisers (PM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) one film-coated tablet of 10 milligram (mg) of BI 1323495 orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal.
- 30 mg BI 1323495 Bid EM: Participants carrying at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) three film-coated tablets of 10 milligram (mg) of BI 1323495 (total dosage=30 mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal.
- 30 mg BI 1323495 Bid PM: Participants carrying no functional allele of the UGT2B17 gene (poor metabolisers (PM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) three film-coated tablets of 10 milligram (mg) of BI 1323495 (total dosage = 30 mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal.
- 70 mg BI 1323495 Bid + Midazolam EM: Participants carrying at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) two film-coated tablets of 10 milligram (mg) and one film-coated tablet of 50 mg of BI 1323495 (total dosage=70 mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal. On Day -1 and on Day 11 participants were also administered a single daily dose of 1.5 mL of solution for injection of midazolam concentrated 50 microgram (ug)/mL (total dosage=75 ug) orally with 240 mL of water within 30 minutes after a standard breakfast.
- 120 mg BI 1323495 Bid + Midazolam EM: Participants with at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) two film-coated tablets of 10 milligram (mg) and two film-coated tablets of 50 mg of BI 1323495 (total dosage=120 mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal. On Day -1 and on Day 11 participants were also administered a single daily dose of 1.5 mL of solution for injection of midazolam concentrated 50 microgram (ug)/mL (total dosage=75 ug) orally with 240 mL of water within 30 minutes after a standard breakfast.
- 120 mg BI 1323495 qd EM: Participants carrying at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 11 once daily (qd) two film-coated tablets of 10 milligram (mg) and two film-coated tablets of 50 mg of BI 1323495 (total dosage=120 mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal.
- 150 mg BI 1323495 Bid + Midazolam EM: Participants carrying at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) one film-coated tablet of 150 milligram (mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal. On Day -1 and on Day 11 participants were also administered a single daily dose of 1.5 mL of solution for injection of midazolam concentrated 50 microgram (ug)/mL (total dosage=75 ug) orally with 240 mL of water within 30 minutes after a standard breakfast.
Period: Overall Study
Arm/Group | Placebo/Placebo + Midazolam | 10 mg BI 1323495 Bid EM | 10 mg BI 1323495 Bid PM | 30 mg BI 1323495 Bid EM | 30 mg BI 1323495 Bid PM | 70 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 qd EM | 150 mg BI 1323495 Bid + Midazolam EM
Started | 22 | 9 | 5 | 9 | 6 | 9 | 9 | 9 | 9
Completed (Not prematurely discontinued trial medication) | 22 | 9 | 5 | 8 | 6 | 8 | 9 | 9 | 8
Not Completed | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The treated set included all subjects who were randomised and treated with at least 1 dose of trial drug. The treatment assignment was determined based on the first treatment the subjects received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Placebo + Midazolam | 10 mg BI 1323495 Bid EM | 10 mg BI 1323495 Bid PM | 30 mg BI 1323495 Bid EM | 30 mg BI 1323495 Bid PM | 70 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 qd EM | 150 mg BI 1323495 Bid + Midazolam EM | Total
Number analyzed (Participants) | 22 | 9 | 5 | 9 | 6 | 9 | 9 | 9 | 9 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.1 (11.1) | 44.3 (15.8) | 36.4 (14.2) | 43.3 (15.4) | 41.2 (15.1) | 44.4 (13.1) | 33.7 (10.3) | 29.9 (9.4) | 35.3 (15.5) | 37.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 4 | 3 | 1 | 4 | 5 | 3 | 3 | 32
  Male | 16 | 6 | 1 | 6 | 5 | 5 | 4 | 6 | 6 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 9 | 5 | 9 | 6 | 9 | 9 | 9 | 9 | 87
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 20 | 9 | 4 | 9 | 6 | 8 | 9 | 9 | 9 | 83
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Drug-related Adverse Events (AEs)
Description: Percentage of participants with treatment-emergent drug-related Adverse Events (AEs) is reported.
  Percentages are calculated using total number of subjects per treatment as the denominator.
Time Frame: Midazolam alone: From administration of midazolam on Day -1 until first administration of BI 1323495 on Day 1, up to 24 hours. All others: From first administration until 7 days after the last administration of BI 1323495, up to 18 days.
Population: Treated Set (TS): The treated set included all subjects who were randomised and treated with at least 1 dose of trial drug. The treatment assignment was determined based on the first treatment the subjects received. Midazolam alone arm consisted of all subjects of the arms "70 mg BI 1323495 bid+Midazolam EM", "120 mg BI 1323495 bid+Midazolam EM", "150 mg BI 1323495 bid+ Midazolam EM" and 9 subjects of the arm "Placebo/Placebo+Midazolam" which were treated with midazolam on Day -1 of the trial.
Measure: Number; unit: percentage of participants
Groups:
- Placebo/Placebo+ Midazolam: This arm comprises placebo only treated participants and those participants who received placebo + midazolam. Placebo only treated participants were administered film-coated tablets of placebo matching BI 1323495 dosage and participants who received placebo + midazolam were administered film-coated tablets of placebo matching BI 1323495 dosage + a single dose of 1.5 ml of solution for injection of midazolam concentrated 50 microgram (ug)/mL (total dosage=75 ug) orally with 240 mL of water within 30 minutes after a standard breakfast on Day -1 and on Day 11.
- Midazolam Alone: This arm consisted of all participants of the arms "70 mg BI 1323495 bid + Midazolam EM", "120 mg BI 1323495 bid + Midazolam EM", "150 mg BI 1323495 bid + Midazolam EM" and 9 subjects of the arm "Placebo/Placebo + Midazolam" which were administered midazolam on Day -1 of the trial. The duration of this analysis phase was approximately 1 day (from Day -1 to first administration of BI 1323495 on Day 1).
- 120 mg BI 1323495 Bid + Midazolam EM: Participants carrying at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) two film-coated tablets of 10 milligram (mg) and two film-coated tablets of 50 mg of BI 1323495 (total dosage=120 mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal. On Day -1 and on Day 11 participants were also administered a single daily dose of 1.5 mL of solution for injection of midazolam concentrated 50 microgram (ug)/mL (total dosage=75 ug) orally with 240 mL of water within 30 minutes after a standard breakfast.
Arm/Group | Placebo/Placebo+ Midazolam | Midazolam Alone | 10 mg BI 1323495 Bid EM | 10 mg BI 1323495 Bid PM | 30 mg BI 1323495 Bid EM | 30 mg BI 1323495 Bid PM | 70 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 qd EM | 150 mg BI 1323495 Bid + Midazolam EM
Number analyzed (Participants) | 22 | 36 | 9 | 5 | 9 | 6 | 9 | 9 | 9 | 9
percentage of participants | 4.5 | 0 | 22.2 | 0 | 33.3 | 16.7 | 11.1 | 22.2 | 0 | 44.4

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 1323495 in Plasma Over a Time Interval of 12 h After Administration of the First Dose (AUC0-12)
Description: Area under the concentration-time curve of BI 1323495 in plasma over a time interval of 12 h after administration of the first dose (AUC0-12) is reported.
Time Frame: Within 3 hours before and 20 minutes (min), 40 min, 1 hour (h), 1.5h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 9h, and 12h after the first administration of BI 1323495 on Day 1.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set included all subjects in the treated set (TS) who provided at least 1 PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if he/she contributed to only 1 PK parameter value for 1 period to the statistical assessment. Only participants with evaluable results for this PK parameter are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours *nanomol/Liter (h*nmol/L)
Groups:
- 70 mg BI 1323495 Bid + Midazolam EM: Participants with at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) two film-coated tablets of 10 milligram (mg) and one film-coated tablet of 50 mg of BI 1323495 (total dosage=70 mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal. On Day -1 and on Day 11 participants were also administered a single daily dose of 1.5 mL of solution for injection of midazolam concentrated 50 microgram (ug)/mL (total dosage=75 ug) orally with 240 mL of water within 30 minutes after a standard breakfast.
- 120 mg BI 1323495 qd EM: Participants with at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 11 once daily (qd) two film-coated tablets of 10 milligram (mg) and two film-coated tablets of 50 mg of BI 1323495 (total dosage=120 mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal.
- 150 mg BI 1323495 Bid + Midazolam EM: Participants with at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) one film-coated tablet of 150 milligram (mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal. On Day -1 and on Day 11 participants were also administered a single daily dose of 1.5 mL of solution for injection of midazolam concentrated 50 microgram (ug)/mL (total dosage=75 ug) orally with 240 mL of water.
Arm/Group | 10 mg BI 1323495 Bid EM | 10 mg BI 1323495 Bid PM | 30 mg BI 1323495 Bid EM | 30 mg BI 1323495 Bid PM | 70 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 qd EM | 150 mg BI 1323495 Bid + Midazolam EM
Number analyzed (Participants) | 9 | 5 | 7 | 6 | 8 | 6 | 9 | 5
hours *nanomol/Liter (h*nmol/L) | 118 (56.1) | 430 (27.2) | 282 (66.2) | 1310 (29.1) | 702 (48.6) | 982 (76.2) | 784 (81.7) | NA (NA) — AUC0-12 could not be calculated due to low number of participants with valid AUC0-12 values.

3. Secondary Outcome: Only for Once Daily (qd) Dosing Group: Area Under the Concentration-time Curve of BI 1323495 in Plasma Over a Uniform Dosing Interval of 24 h After Administration of the First Dose (AUC0-24)
Description: Area under the concentration-time curve of BI 1323495 in plasma over a uniform dosing interval of 24 h after administration of the first dose (AUC0-24) for the once daily (qd) dosing group is reported.
Time Frame: Within 3 hours before and 20 minutes (min), 40 min, 1 hour (h), 1.5h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 9h, 12h and 24 h after administration of BI 1323495 on Day 1.
Population: Pharmacokinetic (PK) parameter analysis set (PKS) of 120 mg BI qd EM arm: This set included all treated subjects of 120 mg BI 1323495 qd EM arm who provided at least 1 PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS of arm, even if he/she contributed to only 1 PK parameter value for 1 period to the statistical assessment. Only participants with evaluable results are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours *nanomol/Liter (h*nmol/L)
Arm/Group | 120 mg BI 1323495 qd EM
Number analyzed (Participants) | 7
hours *nanomol/Liter (h*nmol/L) | 1550 (75.6)

4. Secondary Outcome: Maximum Measured Concentration of BI 1323495 in Plasma After the First Dose (Cmax)
Description: Maximum measured concentration of BI 1323495 in plasma after the first dose (Cmax) is reported.
Time Frame: Within 3 hours before and 20 minutes (min), 40 min, 1 hour (h), 1.5h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 9h, 12h and 24h* after the first administration of BI 1323495 on Day 1. * Applicable only for the 120 mg BI 1323495 qd EM arm.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set included all subjects in the treated set (TS) who provided at least 1 PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if he/she contributed to only 1 PK parameter value for 1 period to the statistical assessment. Only participants with evaluable results of this PK parameter are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/Liter (nmol/L)
Groups:
- 30 mg BI 1323495 Bid EM: Participants with at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) three film-coated tablets of 10 milligram (mg) of BI 1323495 (total dosage=30 mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal.
- 70 mg BI 1323495 Bid + Midazolam EM: Participants with at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) two film-coated tablets of 10 milligram (mg) and one film-coated tablet of 50 mg of BI 1323495 (total dosage=70 mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal. On Day -1 and on Day 11 participants were also administered a single daily dose of 1.5 mL of solution for injection of midazolam concentrated 50 microgram (ug)/mL (total dosage=75 ug) orally with 240 mL of water.
- 120 mg BI 1323495 Bid + Midazolam EM: Participants with at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) two film-coated tablets of 10 milligram (mg) and two film-coated tablets of 50 mg of BI 1323495 (total dosage=120 mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal. On Day -1 and on Day 11 participants were also administered a single daily dose of 1.5 mL of solution for injection of midazolam concentrated 50 microgram (ug)/mL (total dosage=75 ug) orally with 240 mL of water.
Arm/Group | 10 mg BI 1323495 Bid EM | 10 mg BI 1323495 Bid PM | 30 mg BI 1323495 Bid EM | 30 mg BI 1323495 Bid PM | 70 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 qd EM | 150 mg BI 1323495 Bid + Midazolam EM
Number analyzed (Participants) | 9 | 5 | 9 | 6 | 9 | 9 | 9 | 8
nanomol/Liter (nmol/L) | 23.5 (31.4) | 85.3 (30.1) | 62.0 (57.1) | 216 (39.7) | 123 (50.0) | 152 (67.5) | 125 (98.1) | 109 (77.8)

5. Secondary Outcome: Area Under the Concentration-time Curve of BI 1323495 in Plasma at Steady State Over a Uniform Dosing Interval τ (AUCτ,ss)
Description: Area under the concentration-time curve of BI 1323495 in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) is reported. The dosing interval τ is not the same for all groups. The dosing interval is 12 hours (h) for the dose groups with a twice daily (bid) BI 1323495 administration and 24 h for the dose group with a once daily (qd) BI 1323495 administration.
Time Frame: Within 3 hours before and 20 minutes (min), 40 min, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 9h, 12h and 24h* after the last administration of BI 1323495 on Day 11. * Applicable only for the 120 mg BI 1323495 qd EM arm.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours *nanomol/Liter (hnmol/L)
Arm/Group | 10 mg BI 1323495 Bid EM | 10 mg BI 1323495 Bid PM | 30 mg BI 1323495 Bid EM | 30 mg BI 1323495 Bid PM | 70 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 qd EM | 150 mg BI 1323495 Bid + Midazolam EM
Number analyzed (Participants) | 9 | 5 | 8 | 6 | 8 | 9 | 9 | 8
hours *nanomol/Liter (hnmol/L) | 237 (60.8) | 738 (22.8) | 475 (86.2) | 2370 (28.1) | 2490 (59.4) | 2850 (69.4) | 1960 (55.9) | 2070 (41.5)

6. Secondary Outcome: Maximum Measured Concentration of BI 1323495 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmax,ss)
Description: Maximum measured concentration of BI 1323495 in plasma at steady state over a uniform dosing interval τ (Cmax,ss) is reported.
  The dosing interval τ is not the same for all groups. The dosing interval is 12 hours (h) for the dose groups with a twice daily (bid) BI 1323495 administration and 24 h for the dose group with a once daily (qd) BI 1323495 administration.
Time Frame: Within 3 hours before and 20 min, 40 min, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 9h, 12h and 24h* after the last drug administration of BI 1323495 on Day 11. * Applicable only for the 120 mg BI 1323495 qd EM arm.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/liter (nmol/L)
Arm/Group | 10 mg BI 1323495 Bid EM | 10 mg BI 1323495 Bid PM | 30 mg BI 1323495 Bid EM | 30 mg BI 1323495 Bid PM | 70 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 qd EM | 150 mg BI 1323495 Bid + Midazolam EM
Number analyzed (Participants) | 9 | 5 | 8 | 6 | 8 | 9 | 9 | 8
nanomol/liter (nmol/L) | 37.5 (49.6) | 109 (27.7) | 64.4 (78.7) | 300 (32.6) | 281 (48.0) | 362 (77.7) | 164 (48.7) | 265 (46.0)

ADVERSE EVENTS:
Time Frame: Midazolam alone: From administration of midazolam on Day -1 until first administration of BI 1323495 on Day 1, up to 24 hours. All others: From first administration until 7 days after the last administration of BI 1323495, up to 18 days.
Description: Treated Set (TS): The treated set included all subjects who were randomised and treated with at least 1 dose of trial drug. The treatment assignment was determined based on the first treatment the subjects received. Midazolam alone arm consisted of all subjects of the arms "70 mg BI 1323495 bid+Midazolam EM", "120 mg BI 1323495 bid+Midazolam EM", "150 mg BI 1323495 bid+ Midazolam EM" and 9 subjects of the arm "Placebo/Placebo+Midazolam" which were treated with midazolam on Day -1 of the trial.
Groups:
- 70 mg BI 1323495 Bid + Midazolam EM: Participants carrying at least one functional allele of the UGT2B17 gene (extensive metabolisers (EM)) were administered from Day 1 to Day 10 twice daily (bid) and on Day 11 once daily (qd) two film-coated tablets of 10 milligram (mg) and one film-coated tablet of 50 mg of BI 1323495 (total dosage=70 mg) orally with 240 milliliter (mL) of water within 30 minutes (min) of a meal. On Day -1 and on Day 11 participants were also administered a single dose of 1.5 ml of solution for injection of midazolam concentrated 50 microgram (ug)/mL (total dosage=75 ug) orally with 240 mL of water within 30 minutes after a standard breakfast.
Arm/Group | Placebo/Placebo + Midazolam | Midazolam Alone | 10 mg BI 1323495 Bid EM | 10 mg BI 1323495 Bid PM | 30 mg BI 1323495 Bid EM | 30 mg BI 1323495 Bid PM | 70 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 Bid + Midazolam EM | 120 mg BI 1323495 qd EM | 150 mg BI 1323495 Bid + Midazolam EM
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/36 | 0/9 | 0/5 | 0/9 | 0/6 | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/36 | 0/9 | 0/5 | 0/9 | 0/6 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 9/22 | 2/36 | 6/9 | 3/5 | 8/9 | 4/6 | 6/9 | 4/9 | 6/9 | 6/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Placebo + Midazolam (N=22) | Midazolam Alone (N=36) | 10 mg BI 1323495 Bid EM (N=9) | 10 mg BI 1323495 Bid PM (N=5) | 30 mg BI 1323495 Bid EM (N=9) | 30 mg BI 1323495 Bid PM (N=6) | 70 mg BI 1323495 Bid + Midazolam EM (N=9) | 120 mg BI 1323495 Bid + Midazolam EM (N=9) | 120 mg BI 1323495 qd EM (N=9) | 150 mg BI 1323495 Bid + Midazolam EM (N=9)
Headache (Nervous system disorders) | 5 | 2 | 5 | 2 | 6 | 1 | 2 | 2 | 5 | 2
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram PR shortened (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Solar urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laziness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperarousal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tension (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT04107805/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT04107805/SAP_001.pdf